CLINICAL TRIAL: NCT07078305
Title: A Prospective, Single Center, Randomized, Open Label Phase II Clinical Study: Comparing the Combination of Trastuzumab and Regorafenib With Regorafenib Monotherapy for Advanced Hepatocellular Carcinoma After First-line Target Immunotherapy Treatment
Brief Title: Comparing the Combination of Trastuzumab and Regorafenib With Regorafenib Monotherapy for Advanced Hepatocellular Carcinoma After First-line Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E20250415
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; Regorafenib; Tislelizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib; tislelizumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Regorafenib and tislelizumab
- Control group (Active Comparator)
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib and tislelizumab — Tislelizumab: 200mg, iv, d1, Q3W; Regorafenib: 40-120mg, po, qd, d1-21, d22-d28 discontinuation Q4W
  Arms: Experimental group
Drug: Regorafenib — Regorafenib: 40-120mg, po, qd, d1-21, d22-d28 discontinuation Q4W
  Arms: Control group

SUMMARY:
At present, there is no standard treatment plan for hepatocellular carcinoma after the progress of first-line target immunotherapy. Based on the above research background, we believe that the combination of PD-1 inhibitors and multi-target inhibitors is a promising treatment option for second-line liver cancer. Our study aims to explore the efficacy and safety of trastuzumab monoclonal antibody combined with regorafenib compared to regorafenib monotherapy for second-line treatment of advanced hepatocellular carcinoma after previous target immunotherapy progression.

DETAILED DESCRIPTION:
According to GLOBOCAN2020 statistics, in 2020, there were 906000 new cases and 830000 deaths of liver cancer worldwide, making it the seventh most common cancer and the fifth leading cause of cancer death. East Asia, especially China, Japan, and South Korea, is a high-risk area for liver cancer, with China accounting for approximately 50% of the world's new liver cancer cases each year. Epidemiological data show that hepatitis B virus (HBV) infection is the main reason for the high incidence of liver cancer in China. Liver cancer in our country is discovered late and staged late. Most patients have lost the opportunity for surgical resection when they seek medical attention, and the overall prognosis is poor. The 5-year survival rate is about 12.5%.

In recent years, immunotherapy represented by PD-1/PD-L1 inhibitors has continuously brought breakthroughs in the treatment of HCC and has gradually become the cornerstone of advanced liver cancer treatment. The global multicenter Phase III IMbrave150 clinical study compared the combination of atezolizumab and bevacizumab ("T+A" regimen) with sorafenib. The results showed that the overall survival was 19.2 months compared to 13.4 months (HR 0.66, p<0.001), and the progression free survival was 6.9 months compared to 4.3 months (HR 0.65, p<0.001). Compared with sorafenib, the "T+A" regimen significantly improved the overall survival and progression free survival of unresectable HCC patients. In the 194 Chinese patient population, the median OS was 24.0 months compared to 11.4 months (HR 0.53), which is consistent with global benefits. Another randomized, open label, phase II-III ORIENT-32 study showed that the combination of Sintilimab and bevacizumab biosimilar ("Shuangda" regimen) significantly improved patient efficacy compared to sorafenib, significantly reduced the risk of death and progression, improved ORR and quality of life, and subgroup analysis showed similar benefits. The median overall survival of the two groups was 10.4 months (HR=0.569, p<0.001), progression free survival was 4.6 months compared to 2.8 months (HR=0.565, p<0.001), ORR was 21% compared to 4%, and DCR were 72% and 64%, respectively. The combination of Shuangda and each individual drug and potential disease has known safety and good tolerability. Currently, the combination therapy of immune checkpoint inhibitors (anti-PD-1/L1) and anti angiogenic drugs has become the standard treatment for unresectable advanced HCC. Although targeted therapy and immunotherapy have made breakthroughs in the field of liver cancer and continuously extended patient survival, first-line treatment inevitably leads to drug resistance. About 30% of patients cannot achieve objective relief due to primary drug resistance, and the median progression free survival of other patients with first-line treatment is about 4-7 months, followed by secondary drug resistance.

In the second-line treatment of advanced liver cancer, multiple immune monotherapy and anti angiogenic drug monotherapy are recommended by guidelines. The KEYNOTE-394 study enrolled second-line hepatocellular carcinoma (HCC) patients who experienced progression after treatment with sorafenib or oxaliplatin, or were intolerant to sorafenib or oxaliplatin treatment, and randomly assigned them to pembrolizumab+BSC (best supportive treatment) or placebo+BSC. The study results showed that compared with the control group, the pembrolizumab group significantly prolonged the median OS of patients (14.6 months compared to 13.0 months), HR=0.79，P=0.0180）， The 2-year OS rate of the pembrolizumab group was 34.3%, higher than the control group's 24.9%, and the long-term survival benefit was more significant. The median PFS was 2.6 months compared to 2.3 months (HR=0.74, P=0.0032, 2-year PFS rates were 11% and 0%, respectively), and the ORR was 12.7% compared to 1.3%. A global multicenter, randomized, double-blind, placebo-controlled phase III clinical trial of regorafenib in liver cancer patients who had previously received sorafenib treatment showed that after sorafenib treatment, regorafenib significantly reduced the risk of death and disease progression compared to the placebo control group, with a median OS of 10.6 months compared to 7.8 months (HR=0.63, P<0.0001) and a median PFS of 3.1 months compared to 1.5 months (HR=0.46, P<0.0001). However, the above clinical studies included participants who had previously received immunotherapy. In the current situation where target immunotherapy is the mainstream first-line treatment, the recommended plan for second-line treatment is still uncertain. A multicenter real-world study in the Asia Pacific region exploring the progression of first-line treatment with the A+T regimen followed by the selection of second-line system regimens. The median PFS of sorafenib, lenvatinib, and regorafenib were 2.3 months (95% CI 2.0-2.6), 4.0 months (95% CI 3.5-4.9), and 3.6 months (95% CI 2.7-5.4), respectively. The median OS of regorafenib was 6.3 months (95% CI 5.3-7.8), 8.0 months (95% CI 7.0-10.9), and 9.7 months (95% CI 5.2-NR), respectively. The median OS of regorafenib was higher than the other two TKIs. It is worth noting that choosing TKI combined with immune checkpoint inhibitors (IO) as the second-line treatment regimen resulted in higher median PFS and OS than TKI monotherapy, at 5.4 months (95% CI 3.0-8.8) and 12.6 months (95% CI 9.8-NR), respectively.

Although monotherapy immunotherapy or anti angiogenic therapy brings certain benefits to second-line HCC patients, the efficacy is far from meeting clinical needs. Based on the synergistic effect of immunotherapy and anti angiogenic therapy, the combination therapy of the two is also constantly being explored. The JVDJ study showed that the combination of Remdesizumab and Duvalimumab in the treatment of HCC with previous treatment failure had an ORR of 11%, DCR of 61%, median PFS of 4.4 months, and median OS of 10.7 months. The efficacy was better in patients with high PD-L1 expression. A retrospective multicenter study showed that the combination of xindilimab and regorafenib for second-line treatment of advanced liver cancer after first-line sorafenib or lenvatinib treatment resulted in an ORR of 24.1%, DCR of 74.1%, median PFS of 5.6 months, and median OS of 13.4 months.

ELIGIBILITY:
Inclusion Criteria:

* Sign a written informed consent form;
* Age ≥ 18 years old, both male and female are eligible;
* Hepatocellular carcinoma (HCC) diagnosed by organization/pathology or imaging that meets the AASLD diagnostic criteria;
* HCC that has received targeted immunotherapy in the past (regardless of whether local treatment is received or not, excluding neoadjuvant therapy), including atezolizumab+bevacizumab, sintilizumab+bevacizumab analogs, carizolizumab+apatinib, and other PD-1/L1 drugs+TKI, and whose disease progression has been confirmed by imaging;
* Child Pugh score ≤ 7;
* According to RECIST 1.1 criteria, there must be at least one measurable lesion;
* ECOG PS score 0-1;
* Expected survival period greater than 12 weeks;
* The function of important organs meets the following requirements (excluding the use of any blood components and cell growth factors within 14 days):

  1. Blood routine:

     Neutrophils ≥ 1.5 × 109/L Platelet count ≥ 80 × 109/L Hemoglobin ≥ 90g/L;
  2. Liver and kidney function:

Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance rate ≥ 50 ml/min (Cockcroft Gault formula); Total bilirubin (TBIL) ≤ 3 times the upper limit of normal (ULN); AST or ALT levels ≤ 5 times the upper limit of normal (ULN); Urinary protein<2+; If urine protein is ≥ 2+, the 24-hour urine protein quantification must show protein ≤ 1g;

* Normal coagulation function, no active bleeding or thrombotic diseases

  1. International Standardization Ratio INR ≤ 1.5 × ULN;
  2. Partial thromboplastin time APTT ≤ 1.5 × ULN;
  3. Prothrombin time PT ≤ 1.5 × ULN;
* Non surgical sterilization or female patients of childbearing age are required to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill, or condom) during the study treatment period and within 3 months after the end of the study treatment period; Female patients of childbearing age who undergo non-surgical sterilization must have a negative serum or urine HCG test within 7 days prior to enrollment in the study; And it must be during non lactation period; Non surgical sterilization or male patients of childbearing age need to agree to use a medically approved contraceptive measure with their spouse during the study treatment period and within 3 months after the end of the study treatment period.

Exclusion Criteria:

* The subject has previous or concurrent malignant tumors (excluding cured skin basal cell carcinoma and cervical carcinoma in situ);
* It is known that the subject has a history of allergies to large molecule protein preparations, or is known to be allergic to the investigational drug or drug components;
* Within the past 6 months, there have been incidents of esophageal or gastric variceal bleeding caused by portal hypertension; Within 3 months prior to the first administration, severe (G3) varicose veins were identified through endoscopic examination; Evidence of portal hypertension (including imaging findings of splenomegaly), assessed by researchers as high-risk for bleeding
* Any life-threatening bleeding events that have occurred within the past 3 months, including the need for blood transfusion therapy, surgery or local treatment, and continuous medication therapy
* Subjects with any active autoimmune disease or history of autoimmune disease (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, those who have undergone thyroid surgery in the past cannot be included; subjects with vitiligo or complete remission of childhood asthma without any intervention in adulthood can be included; subjects with asthma requiring bronchodilators for medical intervention cannot be included);
* The subject is currently using immunosuppressants, systemic, or absorbable local hormone therapy to achieve immunosuppression (dose>10mg/day prednisone or other therapeutic hormones), and has continued to use it within 2 weeks before enrollment;
* Ascites or pleural effusion with clinical symptoms that require therapeutic puncture or regular drainage (≥ 1 time/month);
* Patients with uncontrolled clinical symptoms or diseases of the heart, such as: (1) NYHA grade 2 or above heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, and (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
* The subject has an active infection or an unexplained fever greater than 38.5 degrees Celsius during the screening period or before the first administration (according to the researcher's judgment, the subject can be included if the fever is caused by the tumor);
* Patients with objective evidence of past and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impairment of lung function, etc;
* Subjects with congenital or acquired immune dysfunction, such as HIV infected individuals;
* Within less than 4 weeks before the study medication, or possibly during the study period, receiving a live vaccine;
* The subject is known to have a history of substance abuse, alcoholism, or drug use;
* Have received Chinese herbal medicine or traditional Chinese patent medicines and simple preparations with anti-tumor indications within 2 weeks before the first administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year
  Progression free survival

SECONDARY OUTCOMES:
ORR | 6 months
  Objective response rate
DCR | 6 months
  Disease Control Rate
OS | 1 year
  Overall survival
AE | 6 months
  Adverse events